CLINICAL TRIAL: NCT04467411
Title: Randomised Controlled Study of Physical Exercise Intervention in Breast Cancer Patients at Risk of Anthracycline-induced Cardiomyopathy:The EMBRACE Study
Brief Title: The EMBRACE Study The EMBRACE Study
Acronym: EMBRACE
Status: Recruiting | Type: Observational
Sponsor: University of Aberdeen (Other)
Responsible Party: Sponsor
Other Study IDs: 2-049-18
Record Dates: First submitted 2020-07-02; First posted 2020-07-13 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples and skeletal muscle biopsies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Breast Cancer Group: Breast Cancer Group
- Healthy Volunteer: Healthy Volunteer Group

SUMMARY:
Cardiomyopathy is a condition that affects the heart muscle, whereby it becomes enlarged, thick or rigid. When the heart muscle becomes involved, it affects the pumping action of the heart. This condition can affect as many as 10% of all patients after undergoing anthracycline cancer drug therapy and unfortunately carries the worst prognosis of all cardiomyopathies. To date, there is no effective intervention that will prevent a patient from developing this condition. The research conducted will look to see if an energy imbalance in the heart predates the onset of detrimental changes to the pumping function of the heart, if this is detected then we can act earlier to prevent the pumping function deteriorating.

DETAILED DESCRIPTION:
There is emerging cellular and experimental evidence that cardiac energetic status is reduced after anthracycline treatment, however, this has not been tested in the human heart. The researchers hypothesize that cardiac energetic status is reduced in the human heart after administration of anthracycline therapy in breast cancer patients, inline with the evidence available from all other types of cardiomyopathies. The researchers propose to use in vivo 31Phosphorus cardiac spectroscopy to measure the cardiac energetic status at the beginning and at the end of the cycles of chemotherapy in the hearts of breast cancer patients who are administered epirubicin (the most modern anthracycline to date) and compare this with the cardiac energetic status of age and gender matched healthy controls. Further, the researchers wish to explore if the myopathy-induced effect of anthracyclines extends to the skeletal muscle as well, by examining skeletal muscle biopsies in these patients.

ELIGIBILITY:
Inclusion Criteria:

* A patient who has been diagnosed with breast cancer and has been scheduled for a first cycle of anthracycline therapy.
* Participant who is willing and able to give informed consent for participation in the study.
* Healthy (gender and age matched) volunteers willing to give informed consent for participation in the study.

Exclusion Criteria:

* Contraindication to magnetic resonance scanning such as an implantable cardiac device.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Only females are eligible to take part in the study
Study Population: Healthy volunteers and patients diagnosed with breast cancer who have been scheduled for the first cycle of anthracycline therapy.
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2030-08-30 (Estimated); Study Completion 2030-08-30 (Estimated)

PRIMARY OUTCOMES:
Cardiac Energetics | At baseline
  Cardiac MRI and MRS
Cardiac Energetics | Through study completion, up to sixteen weeks
  Cardiac MRI and MRS

SECONDARY OUTCOMES:
Cardiac Imaging | At baseline
  Echocardiography
Cardiac Imaging | Through study completion, up to sixteen weeks
  Echocardiography
Blood Biomarkers | At baseline
  BNP and Troponins
Blood Biomarkers | Through study completion, up to sixteen weeks
  BNP and Troponins
Histology | At baseline
  Histology of skeletal muscle biopsies
Histology | Through study completion, up to sixteen weeks
  Histology of skeletal muscle biopsies

CONTACTS AND LOCATIONS:
Overall Officials: Dana Dawson, MD, Principal Investigator — University of Aberdeen
Locations (1):
- Cardiovascular Research Facility, Aberdeen, Aberdeenshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zamorano JL, Lancellotti P, Rodriguez Munoz D, Aboyans V, Asteggiano R, Galderisi M, Habib G, Lenihan DJ, Lip GYH, Lyon AR, Lopez Fernandez T, Mohty D, Piepoli MF, Tamargo J, Torbicki A, Suter TM; ESC Scientific Document Group. 2016 ESC Position Paper on cancer treatments and cardiovascular toxicity developed under the auspices of the ESC Committee for Practice Guidelines: The Task Force for cancer treatments and cardiovascular toxicity of the European Society of Cardiology (ESC). Eur Heart J. 2016 Sep 21;37(36):2768-2801. doi: 10.1093/eurheartj/ehw211. Epub 2016 Aug 26. No abstract available. PMID 27567406
- [Background] Felker GM, Thompson RE, Hare JM, Hruban RH, Clemetson DE, Howard DL, Baughman KL, Kasper EK. Underlying causes and long-term survival in patients with initially unexplained cardiomyopathy. N Engl J Med. 2000 Apr 13;342(15):1077-84. doi: 10.1056/NEJM200004133421502. PMID 10760308
- [Background] Maslov MY, Chacko VP, Hirsch GA, Akki A, Leppo MK, Steenbergen C, Weiss RG. Reduced in vivo high-energy phosphates precede adriamycin-induced cardiac dysfunction. Am J Physiol Heart Circ Physiol. 2010 Aug;299(2):H332-7. doi: 10.1152/ajpheart.00727.2009. Epub 2010 May 21. PMID 20495142
- [Background] Menna P, Salvatorelli E, Minotti G. Anthracycline degradation in cardiomyocytes: a journey to oxidative survival. Chem Res Toxicol. 2010 Jan;23(1):6-10. doi: 10.1021/tx9003424. PMID 19954191
- [Background] Higgins AY, O'Halloran TD, Chang JD. Chemotherapy-induced cardiomyopathy. Heart Fail Rev. 2015 Nov;20(6):721-30. doi: 10.1007/s10741-015-9502-y. PMID 26338137
- [Background] Jones LW, Haykowsky MJ, Swartz JJ, Douglas PS, Mackey JR. Early breast cancer therapy and cardiovascular injury. J Am Coll Cardiol. 2007 Oct 9;50(15):1435-41. doi: 10.1016/j.jacc.2007.06.037. Epub 2007 Sep 24. PMID 17919562
- [Background] Truong J, Yan AT, Cramarossa G, Chan KK. Chemotherapy-induced cardiotoxicity: detection, prevention, and management. Can J Cardiol. 2014 Aug;30(8):869-78. doi: 10.1016/j.cjca.2014.04.029. Epub 2014 May 4. PMID 25064580
- [Background] Kitzman DW, Brubaker PH, Herrington DM, Morgan TM, Stewart KP, Hundley WG, Abdelhamed A, Haykowsky MJ. Effect of endurance exercise training on endothelial function and arterial stiffness in older patients with heart failure and preserved ejection fraction: a randomized, controlled, single-blind trial. J Am Coll Cardiol. 2013 Aug 13;62(7):584-92. doi: 10.1016/j.jacc.2013.04.033. Epub 2013 May 9. PMID 23665370
- [Background] Coats AJ, Adamopoulos S, Radaelli A, McCance A, Meyer TE, Bernardi L, Solda PL, Davey P, Ormerod O, Forfar C, et al. Controlled trial of physical training in chronic heart failure. Exercise performance, hemodynamics, ventilation, and autonomic function. Circulation. 1992 Jun;85(6):2119-31. doi: 10.1161/01.cir.85.6.2119. PMID 1591831
- [Background] O'Connor CM, Whellan DJ, Lee KL, Keteyian SJ, Cooper LS, Ellis SJ, Leifer ES, Kraus WE, Kitzman DW, Blumenthal JA, Rendall DS, Miller NH, Fleg JL, Schulman KA, McKelvie RS, Zannad F, Pina IL; HF-ACTION Investigators. Efficacy and safety of exercise training in patients with chronic heart failure: HF-ACTION randomized controlled trial. JAMA. 2009 Apr 8;301(14):1439-50. doi: 10.1001/jama.2009.454. PMID 19351941
- [Background] Hegde SM, Claggett B, Shah AM, Lewis EF, Anand I, Shah SJ, Sweitzer NK, Fang JC, Pitt B, Pfeffer MA, Solomon SD. Physical Activity and Prognosis in the TOPCAT Trial (Treatment of Preserved Cardiac Function Heart Failure With an Aldosterone Antagonist). Circulation. 2017 Sep 12;136(11):982-992. doi: 10.1161/CIRCULATIONAHA.117.028002. Epub 2017 Jun 21. PMID 28637881
- [Background] Pandey A, Garg S, Khunger M, Darden D, Ayers C, Kumbhani DJ, Mayo HG, de Lemos JA, Berry JD. Dose-Response Relationship Between Physical Activity and Risk of Heart Failure: A Meta-Analysis. Circulation. 2015 Nov 10;132(19):1786-94. doi: 10.1161/CIRCULATIONAHA.115.015853. Epub 2015 Oct 5. PMID 26438781
- [Background] Myers J, Prakash M, Froelicher V, Do D, Partington S, Atwood JE. Exercise capacity and mortality among men referred for exercise testing. N Engl J Med. 2002 Mar 14;346(11):793-801. doi: 10.1056/NEJMoa011858. PMID 11893790
- [Background] Schmitz KH, Courneya KS, Matthews C, Demark-Wahnefried W, Galvao DA, Pinto BM, Irwin ML, Wolin KY, Segal RJ, Lucia A, Schneider CM, von Gruenigen VE, Schwartz AL; American College of Sports Medicine. American College of Sports Medicine roundtable on exercise guidelines for cancer survivors. Med Sci Sports Exerc. 2010 Jul;42(7):1409-26. doi: 10.1249/MSS.0b013e3181e0c112. PMID 20559064
- [Background] Chicco AJ, Schneider CM, Hayward R. Exercise training attenuates acute doxorubicin-induced cardiac dysfunction. J Cardiovasc Pharmacol. 2006 Feb;47(2):182-9. doi: 10.1097/01.fjc.0000199682.43448.2d. PMID 16495754
- [Background] Hydock DS, Wonders KY, Schneider CM, Hayward R. Voluntary wheel running in rats receiving doxorubicin: effects on running activity and cardiac myosin heavy chain. Anticancer Res. 2009 Nov;29(11):4401-7. PMID 20032385
- [Background] Hornsby WE, Douglas PS, West MJ, Kenjale AA, Lane AR, Schwitzer ER, Ray KA, Herndon JE 2nd, Coan A, Gutierrez A, Hornsby KP, Hamilton E, Wilke LG, Kimmick GG, Peppercorn JM, Jones LW. Safety and efficacy of aerobic training in operable breast cancer patients receiving neoadjuvant chemotherapy: a phase II randomized trial. Acta Oncol. 2014 Jan;53(1):65-74. doi: 10.3109/0284186X.2013.781673. Epub 2013 Aug 19. PMID 23957716
- [Background] Jones LW, Liang Y, Pituskin EN, Battaglini CL, Scott JM, Hornsby WE, Haykowsky M. Effect of exercise training on peak oxygen consumption in patients with cancer: a meta-analysis. Oncologist. 2011;16(1):112-20. doi: 10.1634/theoncologist.2010-0197. Epub 2011 Jan 6. PMID 21212429
- [Background] Gouspillou G, Scheede-Bergdahl C, Spendiff S, Vuda M, Meehan B, Mlynarski H, Archer-Lahlou E, Sgarioto N, Purves-Smith FM, Konokhova Y, Rak J, Chevalier S, Taivassalo T, Hepple RT, Jagoe RT. Anthracycline-containing chemotherapy causes long-term impairment of mitochondrial respiration and increased reactive oxygen species release in skeletal muscle. Sci Rep. 2015 Mar 3;5:8717. doi: 10.1038/srep08717. PMID 25732599
- [Background] Octavia Y, Tocchetti CG, Gabrielson KL, Janssens S, Crijns HJ, Moens AL. Doxorubicin-induced cardiomyopathy: from molecular mechanisms to therapeutic strategies. J Mol Cell Cardiol. 2012 Jun;52(6):1213-25. doi: 10.1016/j.yjmcc.2012.03.006. Epub 2012 Mar 21. PMID 22465037
- [Background] Perry CG, Lally J, Holloway GP, Heigenhauser GJ, Bonen A, Spriet LL. Repeated transient mRNA bursts precede increases in transcriptional and mitochondrial proteins during training in human skeletal muscle. J Physiol. 2010 Dec 1;588(Pt 23):4795-810. doi: 10.1113/jphysiol.2010.199448. Epub 2010 Oct 4. PMID 20921196
- [Background] Stephens NA, Gallagher IJ, Rooyackers O, Skipworth RJ, Tan BH, Marstrand T, Ross JA, Guttridge DC, Lundell L, Fearon KC, Timmons JA. Using transcriptomics to identify and validate novel biomarkers of human skeletal muscle cancer cachexia. Genome Med. 2010 Jan 15;2(1):1. doi: 10.1186/gm122. PMID 20193046
- [Background] Barwell ND, Malkova D, Moran CN, Cleland SJ, Packard CJ, Zammit VA, Gill JM. Exercise training has greater effects on insulin sensitivity in daughters of patients with type 2 diabetes than in women with no family history of diabetes. Diabetologia. 2008 Oct;51(10):1912-9. doi: 10.1007/s00125-008-1097-6. Epub 2008 Jul 29. PMID 18663427
- [Background] Dawson DK, Neil CJ, Henning A, Cameron D, Jagpal B, Bruce M, Horowitz J, Frenneaux MP. Tako-Tsubo Cardiomyopathy: A Heart Stressed Out of Energy? JACC Cardiovasc Imaging. 2015 Aug;8(8):985-7. doi: 10.1016/j.jcmg.2014.10.004. Epub 2014 Nov 1. No abstract available. PMID 25499134
- [Background] Naressi A, Couturier C, Castang I, de Beer R, Graveron-Demilly D. Java-based graphical user interface for MRUI, a software package for quantitation of in vivo/medical magnetic resonance spectroscopy signals. Comput Biol Med. 2001 Jul;31(4):269-86. doi: 10.1016/s0010-4825(01)00006-3. PMID 11334636
- [Derived] Gamble DT, Ross J, Khan H, Unger A, Cheyne L, Rudd A, Saunders F, Srivanasan J, Kamya S, Horgan G, Hannah A, Baliga S, Tocchetti CG, Urquhart G, Linke WA, Masannat Y, Mustafa A, Fuller M, Elsberger B, Sharma R, Dawson D. Impaired Cardiac and Skeletal Muscle Energetics Following Anthracycline Therapy for Breast Cancer. Circ Cardiovasc Imaging. 2023 Oct;16(10):e015782. doi: 10.1161/CIRCIMAGING.123.015782. Epub 2023 Oct 17. PMID 37847761